CLINICAL TRIAL: NCT03869385
Title: Randomised Controlled Multicentre Study of Albumin Replacement Therapy in Septic Shock
Brief Title: Albumin Replacement Therapy in Septic Shock
Acronym: ARISS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sustained low inclusion rates.
Sponsor: Jena University Hospital (Other)
Collaborators: German Research Foundation (Other); Instituto Grifols, S.A. (Industry); University Hospital Goettingen (Other); SepNet - Critical Care Trials Group (Other); Center for Sepsis Control and Care, Germany (Other)
Responsible Party: Principal Investigator, Yasser Sakr, Prof. Dr., Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZKSJ0112_ARISS; 2018-001874-89 (EudraCT Number); SA 2167/3-1, Nr: 328809707 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG)); ZKSJ0112 (Other: Trial code, ZKS Jena)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock
Keywords: Human albumin; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Albumins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Albumin group (Experimental): Patients assigned to the Albumin group will receive a 60 g loading dose of human albumin 20% over 2-3 hours. Serum albumin levels will be maintained at least at 30 g/l in the ICU for a maximum of 28 days following randomization using 40-80 g human albumin 20% infusion.
  Interventions: Drug: Albutein® 200 g/L or Plasbumin® 20
- Control group without albumin: (No Intervention): The control group will be treated according to the usual practice with crystalloids as the first choice for the resuscitation and maintenance phase of septic shock.

INTERVENTIONS:
Drug: Albutein® 200 g/L or Plasbumin® 20 — The initial dose of the trial drug must be started within 6 to 24 hours after the beginning of the septic shock. Starting dose: 60 g human albumin 20% (Albutein® 200 g/L, infusion solution) over 2-3 h Daily administration of the trial drug will be based on the serum albumin concentration measured each day. Dose adjustment will follow a predetermined schedule with the aim of maintaining a serum albumin concentration of at least 30 g/l. Administration of the trial drug will continue for a maximum of 28 study days after randomisation and only as long as the participant is being treated in the ICU.
  Other Names: Human Albumin 20%
  Arms: Albumin group

SUMMARY:
Albumin is a key regulator of fluid distribution within the extracellular space and possesses several properties beyond its oncotic activity, including binding and transport of several endogenous molecules, anti-inflammatory and anti-oxidant actions, nitric oxide modulation, and buffer function. The accumulating evidence suggests that supplementation of albumin may provide survival advantages only when the insult is severe as in patients with septic shock. Prospective randomized trials on the possible impact of albumin replacement in these patients with septic shock are lacking. The aim of the study is to investigate whether the replacement with albumin and the maintenance of its serum levels at least at 30 g/l for 28 days improve survival in patients with septic shock compared to resuscitation and volume maintenance without albumin. In this prospective, multicenter, randomised trial, adult patients (≥18 years) with septic shock will be randomly assigned within a maximum of 24 hours after the onset of septic shock after obtaining informed consents to treatment or control groups. Patients assigned to the treatment group will receive a 60 g loading dose of human albumin 20% over 2-3 hours. Serum albumin levels will be maintained at least at 30 g/l in the ICU for a maximum of 28 days following randomization using 40-80 g human albumin 20% infusion. The control group will be treated according to the usual practice with crystalloids as the first choice for the resuscitation and maintenance phase of septic shock. The primary end point is 90 days mortality and secondary end points include 28-day, 60-day, ICU, and in-hospital mortality, organ dysfunction/failure, and length of ICU and hospital stay. In total 1412 patients need to be analyzed, 706 per group. Assuming a dropout rate of 15%, a total of 1662 patients need to be allocated.

DETAILED DESCRIPTION:
This is a prospective, multicentre, randomised, controlled, parallel-grouped, open-label, interventional clinical trial in which 1662 patients are planned to be allocated. Subjects will be randomized in a 1:1 ratio to receive either Albumin or routine treatment with crystalloids. Treatment will be continued at maximum for 28 days or until the patient leaves the ICU. Primary endpoint measurement will be carried out 90 days after randomisation

ELIGIBILITY:
Inclusion Criteria:

* The presence of septic shock meeting all of the following criteria:

  * Clinically possible or probable or microbiologically confirmed infection taking into account the definitions of the "International Sepsis Forum (ISF)"
  * Despite adequate volume therapy, vasopressors are required to maintain mean arterial pressure (MAP) ≥ 65 mm Hg for at least 1 hour
  * Serum lactate level > 2 mmol/l (18 mg/dl) despite adequate volume therapy
* Start of septic shock less than 24 hours prior to inclusion, so that the start dose of the trial drug in the albumin group will be possible within 6-24 hours after the start of the septic shock
* Age: ≥ 18 years
* Written informed consent of the patient or his/her legal representative or confirmation of the urgency of participation in the clinical trial and possible benefit to the patient by an independent consultant or the implementation of other established procedures according to the local regulations of the contributing centre to include patients who are unable to provide informed consent in whom subsequent consent may be obtained retrospectively.
* Patients of childbearing age: negative pregnancy test

Exclusion Criteria:

* Moribund conditions with life expectancy less than 28 days because of comorbid conditions or advanced malignant disease and palliative situations with life expectancy less than 6 months
* Presence of an "end of life" decision prior to obtaining informed consent: "Do Not Resuscitate (DNR)" and "Withhold/Withdraw Life-Sustaining measures"
* Previous participation in this study
* Participation in another interventional clinical trial within the past 3 months
* Shock states that can be explained by other causes, e.g. cardiogenic shock, anaphylactic shock, neurogenic shock
* History of hypersensitivity to albumin or any other component of the trial drug, e.g., B., sodium caprylate, sodium N-acetyltryptophanate
* Diseases in which albumin administration may be deleterious, e.g., decompensated heart failure or traumatic brain injury
* Clinical conditions where albumin administration is indicated, e.g., hepatorenal syndrome, nephrosis, burns, intestinal malabsorption syndrome
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Sakr, MD, PhD, Principal Investigator — Jena University Hospital
Locations (27):
- Germany (27):
  - Klinikum Augsburg, Klinik für Anästhesiologie und Operative Intensivmedizin, Augsburg
  - Helios Klinikum Bad Saarow, Klinik für Intensivmedizin, Bad Saarow
  - Vivantes Humboldt Klinikum, Klinik für Innere Medizin, Kardiologie und konservative Intensivmedizin, Berlin
  - Universitätsklinikum Bonn, Klinik für Anästesiologie und Operative Intensivmedizin, Bonn
  - St. Elisabeth Krankenhaus, Klinik für Anästhesiologie, Operative Intensivmedizin und Schmerztherapie, Cologne
  - Universitätsklinikum Erlangen, Anästesiologische Klinik, Erlangen
  - Universitätsklinikum Freiburg, Klinik für Allgemein- und Viszeralchirurgie, Chir. Intensivstation, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Klinik für Anästhesiologie, Rettungs- und Intensivmedizin, Göttingen
  - Universitätsmedizin Greifswald, Klinik für Anästhesiologie, Intensiv-, Notfall- und Schmerzmedizin, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Intensivmedizin, Hamburg
  - Universitätsklinikum Heidelberg, Klinik für Anästhesiologie, Heidelberg
  - Klinikum Herford, Medizinische Klinik III, Kardiologie, Herford
  - Marien Hospital Herne, Universitätsklinikum der Ruhr-Universität Bochum, Klinik für Anästhesiologie, Operative Intensivmedizin, Schmerztherapie, Palliativmedizin, Herne
  - Universitätsklinikum des Saarlandes, Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Homburg
  - Universitätsklinikum Jena, Innere Medizin I, Kardiologie, Jena
  - Universitätsklinikum Jena, Klinik für Innere Medizin I, Kardiologie, Jena
  - Universitätsklinikum Schleswig-Holstein, Klinik für Operative Intensivmedizin, Kiel
  - Universitätsklinikum Leipzig, Interdisziplinäre Internistische Intensivmedizin, Leipzig
  - Universitätsklinikum Leipzig, Klinik für Anästhesiologie u. Intensivtherapie, Leipzig
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Neurologie, Leipzig
  - Universitätsklinikum Magdeburg, Klinik für Innere Medizin, Kardiologie und Angiologie, Magdeburg
  - Universitätsklinikum Magdeburg, Klinik für Anästhesiologie und Intensivmedizin, Magdeburg
  - Universitätsklinikum der Johannes-Gutenberg-Universität Mainz, Klinik für Anästhesiologie, Mainz
  - Klinikum der LMU München, Klinik für Anästhesiologie, München
  - Klinikum rechts der Isar der TU München, Klinik für Anästhesiologie und Intensivmedizin, München
  - Universitätsklinikum Münster, Klinik für Anästesiologie, operative Intensivmedizin und Schmerztherapie, Münster
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Chirurgie, Regensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakr Y, Bauer M, Nierhaus A, Kluge S, Schumacher U, Putensen C, Fichtner F, Petros S, Scheer C, Jaschinski U, Tanev I, Jacob D, Weiler N, Schulze PC, Fiedler F, Kapfer B, Brunkhorst F, Lautenschlaeger I, Wartenberg K, Utzolino S, Briegel J, Moerer O, Bischoff P, Zarbock A, Quintel M, Gattinoni L; SepNet - Critical Care Trials Group. Randomized controlled multicentre study of albumin replacement therapy in septic shock (ARISS): protocol for a randomized controlled trial. Trials. 2020 Dec 7;21(1):1002. doi: 10.1186/s13063-020-04921-y. PMID 33287911

RESULTS

PARTICIPANT FLOW:
Groups:
- Albumin Group: Patients assigned to the Albumin group received a 60 g loading dose of human albumin 20% over 2-3 hours. Serum albumin levels were maintained at least at 30 g/l in the ICU for a maximum of 28 days following randomization using 40-80 g human albumin 20% infusion.
- Control Group Without Albumin:: The control group was treated according to the usual practice with crystalloids as the first choice for the resuscitation and maintenance phase of septic shock.
Period: Overall Study
Arm/Group | Albumin Group | Control Group Without Albumin:
Started | 222 | 218
Completed | 222 | 218
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Informed consents were not possible to obtain within 72 hours after randomization in 14 patients, 4 patients were lost to follow up, 2 patients withdrew the informed consent, and the study was terminated in one patient due to investigator decision. Therefore, the primary outcome parameter was available for analysis in 210 patients in the albumin and 209 patients in the control groups
Groups:
- Control Group Without Albumin:: The control group was treated according to the usual practice with crystalloids as the first choice for the resuscitation and maintenance phase of septic shock.
  The demographic and baseline characteristics were similar between the study groups.
- Total: Total of all reporting groups
Arm/Group | Albumin Group | Control Group Without Albumin: | Total
Number analyzed (Participants) | 222 | 218 | 440
Age, Continuous [Median (Full Range); unit: years] | 69.5 [29 to 89] | 68.5 [23 to 87] | 69 [23 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 70 | 150
  Male | 142 | 148 | 290
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 222 | 218 | 440
Blood lactate level [Median (Inter-Quartile Range); unit: mmol/liter] | 4.9 [4.4 to 5.3] | 5 [4.3 to 5.6] | 4.9 [4.4 to 5.5]
Serum albumin [Mean (Standard Deviation); unit: g/liter] | 22 (6) | 22 (6) | 22 (6)

OUTCOME MEASURES:

1. Primary Outcome: 90-day All Cause Mortality
Description: Mortality within 90 days after randomisation
Time Frame: 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 210 | 209
Participants | 91 | 96

2. Secondary Outcome: 28-day Mortality
Description: Mortality within 28 days after randomisation
Time Frame: 28 days
Population: At 28 days after randomization, informed consent was not possible to be obtained within 72 hours of randomization in 14 patients, 2 patients withdrew consent, and the study was terminated in one patient due to investigator decision. Therefore, 28-days mortality were available in 213 vs. 210 patients in the albumin vs. control group, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 213 | 210
Participants | 66 | 80

3. Secondary Outcome: 60-day Mortality
Description: Mortality within 60 days after randomisation
Time Frame: 60 days
Population: At 60 days after randomization, informed consent was not possible to be obtained within 72 hours of randomization in 14 patients, 2 patients withdrew consent, 2 patients were lost to follow-up, and the study was terminated in one patient due to investigator decision. Therefore, 60-days mortality were available in 211 vs. 210 patients in the albumin vs. control group, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 211 | 210
Participants | 82 | 95

4. Secondary Outcome: Organ Failure
Description: Organ failure defined as increase in the daily recorded Sequential organ Failure Assessement (SOFA) subscores; cardiovascular, respiratory, hematologic, hepatic, renal, neurologic (range 0-4 points each) from a value <2 to a value ≥ 2
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
participants
  1 organ failure | 68 | 52
  2 organ failures | 19 | 14
  3 organ failures | 2 | 7
  4 organ failures | 0 | 1

5. Secondary Outcome: Sequential Organ Failure Assessement (SOFA) Score
Description: The overall degree of organ dysfunction/failure assessed daily by the total Sequential Organ Failure Score (SOFA score: range 0-24 points), with higher scores indicating higher degree of overall organ dysfunction/failure).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
Points | 9 (0.5) | 8.6 (0.7)

6. Secondary Outcome: ICU Length of Stay
Description: Intensive Care unit stay of first hospitalization after randomisation within 90 days
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
Days | 13 [7 to 22] | 12 [7 to 29]

7. Secondary Outcome: Hospital Length of Stay
Description: Hospital stay of first hospitalization after randomisation within 90 days
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
Days | 24 [15 to 42] | 27 [14 to 45]

8. Secondary Outcome: Ventilation-free Days
Description: Ventilation-free days within 28 days after randomisation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
Days | 4 [1 to 7] | 3 [0 to 7]

9. Secondary Outcome: Vasopressor-free Days
Description: Vasopressor-free days within 28 days after randomisation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
Days | 2.5 [0 to 7] | 2 [0 to 6]

10. Secondary Outcome: Total Amount of Fluid of Fluid Administration and Total Fluid Balance in the ICU.
Description: Total amount of fluid of fluid administration and total fluid balance in the ICU within 28 days after randomisation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: ml/day
Arm/Group | Albumin Group | Control Group Without Albumin:
Number analyzed (Participants) | 222 | 218
ml/day
  Total amount of fluid adminstration | 3200 [2502 to 3544] | 3693 [2540 to 4443]
  Total fluid balance | 234 [-491 to 1290] | 355 [-402 to 1576]

ADVERSE EVENTS:
Time Frame: In the albumin group until 24 h after the last dose of the trial drug Iin the control group without albumin until day 28 after randomisation or until discharge from the ICU, if it occurs before day 28 after randomisation. In the event that adverse events are still "ongoing" after the above dates, they were tracked until maximum the end of data collection (Day 90). If they are "ongoing" on day 90, they were documented as "not recovered," "recovered with sequelae," or "unknown."
Description: Events plausibly explainable by sepsis were recorded in both groups as sepsis-related clinical events, but not as adverse events (AEs). Documentation of the sepsis-related clinical event as an AE occurs only if the examiner suspects a connection with the administration of the trial drug, which is therefore only possible in the albumin group. Clinically relevant worsening of a pre-existing disease not related to sepsis was considered and documented as an AE.
Arm/Group | Albumin Group | Control Group Without Albumin:
All-Cause Mortality (participants affected / at risk) | 91/222 | 96/218
Serious Adverse Events (participants affected / at risk) | 3/222 | 2/218
Other Adverse Events (participants affected / at risk) | 183/222 | 176/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin Group (N=222) | Control Group Without Albumin: (N=218)
Hypervolemia (Cardiac disorders) | 3 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin Group (N=222) | Control Group Without Albumin: (N=218)
Sepsis related, Cardiovascular events (Vascular disorders) | 183 | 176

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03869385/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT03869385/SAP_003.pdf